CLINICAL TRIAL: NCT06334289
Title: A Predictive Study of Peripheral Blood Biomarkers on Postoperative Neurocognitive Dysfunction in Elderly Frail and Non-frail Patients Undergoing Gastrointestinal Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Yongtao Sun, professor, Qianfoshan Hospital
Other Study IDs: YXLL-KY-2024(017)
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Perioperative Neurocognitive Disorders; Frail Elderly
Keywords: Peripheral blood biomarkers; inflammatory markers; Alanine aminotransferase; blood lipids; vitamin D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frailty group
- Non-frailty group

SUMMARY:
Perioperative neurocognitive impairment (PND) mainly includes acute postoperative delirium (POD) and persistent postoperative cognitive impairment (POCD), which are common postoperative complications in elderly patients. Perioperative neurocognitive impairment (PND) is attracting increasing attention, but its exact mechanism is still unclear. The diagnosis of PND lacks the gold standard, so it is difficult to determine the incidence rate. At present, the diagnosis is mainly conducted through the scale. Therefore, this study aims to explore the correlation between peripheral blood biomarkers and PND in elderly frail patients undergoing gastrointestinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old
* American Society of Anesthesiologists (ASA) classification: grades I-IV
* Hospitalization time ≥ 3 days

Exclusion Criteria:

* The revised version of the Cognitive Function Telephone Questionnaire (TICS-M) was used before surgery to determine cognitive impairment (TICS-M score ≤ 27 points)
* Refuse to participate
* Emergency surgical patients
* Central nervous system diseases (dementia, depression, etc.)
* Severe renal insufficiency (requiring dialysis)
* Long term use of psychotropic drugs (such as clozapine, risperidone, olanzapine, haloperidol, chlorpromazine, etc.)
* History of alcohol abuse or use of acetylcholine drugs
* The same patient can only be included once, regardless of whether the reason for the second surgery is related to the first cause

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients undergoing gastrointestinal surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 338 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative 7-day incidence of PND | 30 days after surgery
  The primary outcome of this study is the postoperative 7-day incidence of PND Blood samples (approximately 3ml each time) were taken before anesthesia induction and after the removal of the tracheal catheter, and then standardized tests were performed to analyze the blood markers related to this study. The follow-up method used was the revised version of the Cognitive Function Telephone Questionnaire (TICS-M), and the scores were evaluated through telephone follow-up. Screening was conducted one day before surgery, and follow-up and diagnosis were conducted on the 7th and 30th days after surgery. When the reliable change index of TICS-M score decreases by 1-2, POCD is considered mild. When the reliable change index of TICS-M score decreases by ≥ 2, POCD is considered severe. After follow-up, the values of serum biomarkers were obtained from two groups of patients for data analysis, and the correlation between the biomarkers and the two groups was obtained.